CLINICAL TRIAL: NCT06174194
Title: Effect of Sugar-Free Chewing Gum Containing Tulsi Extract on Salivary Streptococcus Mutans in a Group of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Somaya Mohsena Anwar, Pediatric Dentist, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REC-PE-23-14
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dental Caries in Children
Keywords: caries prevention; streptococcus mutans

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tulsi Gum Arm (Experimental): All participants were instructed to masticate gum containing Tulsi extract for a duration of 5 minutes and subsequently discard the gum. Salivary samples were collected before commencing gum chewing and after 30 minutes following the conclusion of chewing gum for 5 minutes.
  Interventions: Dietary Supplement: Tulsi Gum

INTERVENTIONS:
Dietary Supplement: Tulsi Gum — The intervention involves participants chewing a specially formulated gum known as "Tulsi Gum" for 5 minutes. Tulsi Gum contains Tulsi extract, a natural substance derived from the Tulsi plant. This extract is recognized for its potential antimicrobial properties. Participants are then required to discard the gum. The study aims to assess the effect of Tulsi Gum on salivary Streptococcus mutans count in children aged 4 to 11 years. This assessment contributes to understanding the potential of Tulsi Gum in preventing dental caries in children.

SUMMARY:
The goal of this clinical trial was to explore how adding Tulsi extract, a natural plant substance, to chewing gum affects the levels of Streptococcus mutans, type of bacteria that cause dental caries, in the saliva of children aged 4 to 11 years. Participants should not use removable prosthetics or orthodontic appliances and had had not used antibiotics in the 2 weeks preceding sample collection.

We want to answer this main question:

Can chewing gum with Tulsi extract significantly reduce the number of Streptococcus mutans bacteria in children's saliva?

Participants tasks:

* Children were asked to chew gum containing Tulsi extract for 5 minutes and then dispose of the gum.
* Two salivary samples were collected from each child: one before gum chewing and another 30 minutes after disposing the gum.

Researchers compared Streptococcus mutans counts in saliva before and after gum chewing to determine if there is a significant reduction in bacterial colonies.

DETAILED DESCRIPTION:
This interventional clinical trial aimed to assess the antimicrobial effect of Tulsi extract incorporated into chewing gum on the salivary Streptococcus mutans count in a group of children aged 4 to 11 years. The study enrolled 32 systemically healthy children who met specific criteria, including the absence of removable prosthetics or orthodontic appliances and no recent history of antibiotic use in the preceding 2 weeks.

Participants and Methods:

A sample of 33 children within the age range of 4 to 11 years was selected. The participants were systemically healthy, without removable prosthetics or orthodontic appliances, and had no recent history of antibiotic use in the previous 2 weeks. To standardize saliva collection conditions, samples were collected between 9-10 am in the morning. Children were instructed not to eat or drink anything (except water) 1 hour before saliva collection to maintain consistency in the samples.

Participants were then asked to spit into sterile containers as the method of saliva collection. Subsequently, they were instructed to masticate gum containing Tulsi extract for a duration of 5 minutes and discard the gum.

Two salivary samples were collected from each participant: one before commencing gum chewing and another 30 minutes after the conclusion of chewing gum for 5 minutes. The samples were streaked onto mitis salivarius agar plates and incubated at 37°C for 24 hours. Streptococcus mutans colonies were then counted to assess the change in bacterial count.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 4 and 12 years old.
2. No fixed or removable orthodontic appliances or removable prostheses.
3. Systemically healthy patients.
4. No history of recent antibiotic administration (previous 2 weeks).

Exclusion Criteria:

1. History of using antimicrobial mouthwash (previous 12 hours).
2. History of fluoride treatment (previous 2 weeks).

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Salivary Streptococcus mutans Count | Assessment will be conducted at two specific time points for each participant: Before commencing gum chewing, and after 30 minutes following the conclusion of chewing Tulsi Gum for 5 minutes...
  The primary outcome measure involves assessing the count of Streptococcus mutans colonies in salivary samples. This count serves as a metric for evaluating the antimicrobial effect of Tulsi Gum on dental caries prevention in children.

CONTACTS AND LOCATIONS:
Overall Officials: somaya MA Kahwa, Dr, Principal Investigator — Faculty of Dental Medicine for Girls
Locations (1):
- Faculty of Dental Medicine Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No